CLINICAL TRIAL: NCT03282318
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Parallel-group, Proof of Concept Study to Investigate Efficacy, Safety, Pharmacodynamics and Pharmacokinetics of ASP6294 in the Treatment of Female Subjects With Bladder Pain Syndrome/Interstitial Cystitis
Brief Title: A Study to Investigate Efficacy, Safety, Pharmacodynamics and Pharmacokinetics of ASP6294 in the Treatment of Female Subjects With Bladder Pain Syndrome/Interstitial Cystitis
Acronym: SERENITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6294-CL-0101; 2016-004138-12 (EudraCT Number)
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Bladder Pain Syndrome; Interstitial Cystitis
Keywords: Bladder Pain Syndrome; Interstitial Cystitis; ASP6294
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASP6294 (Experimental): Participants will receive 320 mg ASP6294 subcutaneous injection at 4-week intervals at baseline (Day 1/Week 0), Week 4 and Week 8.
  Interventions: Drug: ASP6294
- Placebo (Placebo Comparator): Participants will receive placebo to match 320 mg ASP6294 subcutaneous injection at 4-week intervals at baseline (Day 1/Week 0), Week 4 and Week 8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP6294 — Participants will receive 320 mg ASP6294 subcutaneous injection at 4-week intervals at baseline (Day 1/Week 0), Week 4 and Week 8.
  Arms: ASP6294
Drug: Placebo — Participants will receive placebo to match 320 mg ASP6294 subcutaneous injection at 4-week intervals at baseline (Day 1/Week 0), Week 4 and Week 8.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate efficacy, safety and tolerability of ASP6294 in female participants with Bladder Pain Syndrome/Interstitial Cystitis (BPS/IC). This study will also investigate the pharmacokinetics (PK) and pharmacodynamics (PD) of ASP6294 in female participants with BPS/IC.

ELIGIBILITY:
Inclusion Criteria:

* Subject's signs, symptoms and diagnostic work-up are in accordance with the international society for the study of bladder pain syndrome (ESSIC) definition for bladder pain syndrome/interstitial cystitis (BPS/IC): pelvic pain, pressure or discomfort perceived to be related to the urinary bladder accompanied by at least 1 other urinary symptom such as persistent urge to void or frequency, for at least 6 months in absence of urinary infection or other obvious pathology or identifiable causes. There is documented proof of the diagnosis BPS/IC that has been entered into the subject's records at least 2 months prior to Visit 1/Screening.
* Subject has a score of ≥ 4 and ≤ 9 for pain as assessed by scoring the average pain of the week preceding Visit 1/Screening, using an 11-point NRS (0-10).
* Subject has an estimated voiding frequency of ≥ 8 and ≤ 30 voids per 24 hours.
* Subject has a score of ≥ 7 on the interstitial cystitis symptom index (ICSI) questionnaire.
* Subject must either:

  * Be of nonchildbearing potential:
  * Postmenopausal (defined as at least 1 year without any menses for which there is no other obvious pathological or physiological cause) prior to screening, or
  * Documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy)
  * Or, if of childbearing potential,
  * Agree not to try to become pregnant during the study and for 5 half-lives (i.e., 70 days) after the final study drug administration at Visit 5/Week 8, and
  * Have a negative urine pregnancy test at Visit 1/Screening, and
  * If heterosexually active, agree to consistently use 1 form of highly effective birth control starting at screening and throughout the study period and for 5 half-lives (i.e., 70 days) after the final study drug administration at Visit 5/Week 8.
* Subject must agree not to breastfeed starting at screening and throughout the study period, and for 5 half-lives (i.e., 70 days) after the final study drug administration at Visit 5/Week 8.
* Subject must agree not to donate ova starting at screening and throughout the study period, and for 5 half-lives (i.e., 70 days) after the final study drug administration at Visit 5/Week 8.
* Subject must be willing and able to comply with study requirements (e.g., complete questionnaires and diaries, able to read and attend all required study visits).
* Subject agrees not to participate in another interventional study while participating in the present study (i.e., between Visit 1/Screening and Visit 7/Week 18).
* Subject has undergone at least 2 different therapies for BPS/IC with unsatisfactory results, prior to study entry.
* Subject has at least moderate pain as reflected by an average MDP of ≥ 4.0 and ≤ 9.0. The average MDP is the average of daily assessments of MDP in the week prior to the visit with at least 5 recordings. Additionally, the MDP recordings must not differ over 4 points between consecutive days.
* Subject has a mean voiding frequency of ≥ 8.0 and ≤ 30.0 per 24 hours as assessed with the 3 day electronic micturition diary in the week prior to the visit.
* Subject is confirmed to be willing to comply and has shown to be compliant with all study requirements during the run-in period.

Exclusion Criteria:

* Subject has osteoarthritis or has a history of rapidly progressive osteoarthritis.
* Subject has a score of ≥ 30 on the Pain Catastrophizing Scale (PCS).
* Subject has a score of > 12 on the HADS-D (Hospital Anxiety and Depression Scale - Depression subscale).
* Subject has significant pelvic floor pain or spasm which is considered the main cause of the chronic pelvic/bladder pain as concluded by the investigator based on the pelvic floor examination.
* Subject has undergone a fulguration or excision of a Hunner's lesion any time prior to the screening visit.
* Subject has recently undergone or started treatment for BPS/IC as specified below:

  * subject has undergone a cystoscopy with hydrodistension or Botox injections in the bladder within 6 months prior to the screening visit.
  * subject has received non-pharmacological interventions for BPS/IC (including but not limited to electric stimulation therapy or acupuncture therapy) within 3 months prior to the screening visit.
  * subject has received any intravesical pharmacological treatment for BPS/IC (including but not limited to heparin or dimethyl sulfoxide) within 4 weeks prior to the screening visit
  * subject had an initiation, discontinuation, or variation in the dose and/or frequency of antimuscarinics, mirabegron, antidepressants (including amitriptyline), anticonvulsants, benzodiazepines, skeletal muscle relaxants, nonsteroidal anti-inflammatory drugs, non-opioid analgesics, pentosan polysulphate sodium, homeopathic medication and/or herbal therapies during the last 4 weeks prior to the screening visit.
  * subject has had changes in non-pharmacological treatment for BPS/IC (e.g., diet or physical therapy) during the last 4 weeks prior to the screening visit.
* Subject has bladder pathology as specified below:

  * a post-void residual (PVR) >200 mL.
  * subject has a known currently symptomatic urethral diverticulum.
  * subject has genital tract condition or pelvic pathology (e.g., post-partum, post-pelvic surgery, post-hysterectomy) that may complicate diagnosis and the evaluation of pelvic pain and urinary symptoms. Note: A history of a Cesarean section is not a reason for exclusion.
  * subject has a known currently symptomatic bladder or ureteral calculi.
  * subject currently has cystitis (radiation cystitis, Bacillus Calmette-Guérin-induced cystitis, bacterial/tuberculous cystitis, cyclophosphamide cystitis) or has had a documented symptomatic bacterial cystitis within the last 1 month prior to the screening visit. In case of bacterial cystitis (UTI), the subject can be re-screened 1 month after successful treatment.
  * subject has currently clinically significant urinary bladder abnormalities (e.g., bladder mass, bladder stone, bladder diverticulum, small contracted end-stage bladder), except for abnormalities associated with BPS/IC.
  * subject has had any invasive procedures of either the urinary bladder, urethra, ureter or renal pelvis (e.g., transurethral resection of bladder [including bladder biopsy], urethral dilatation, endovesicular lithotripsy) within 3 months prior to the screening visit.
  * subject has a known current neurologic disease or a defect affecting urinary bladder function (e.g., neurogenic bladder, systemic or central neurological disease, such as Multiple Sclerosis or Parkinson's disease).
  * subject has a known current lower urinary tract malignancy. In case of positive sediment (micro) hematuria results, local procedures/guidelines will need to be followed to exclude malignancy. Only if hematuria has been present within the last 6 months and malignancy has been adequately ruled out by the investigator according to local diagnostic procedures, the subject does not have to be excluded. Note that if the subject had a (negative) bladder biopsy, the subject can only be re-screened after 3 months following this biopsy. Documentation of all diagnostic outcomes and investigator's decisions need to be available.
* Subject has a known history of, or currently has inflammatory bowel disease (i.e., Crohn's Disease or Ulcerative Colitis) and/or Sjögren Syndrome.
* Subject has a known current severe constipation and/or severe diarrhea, severe active diverticulitis and/or severe gastrointestinal bleeding.
* Subject has a known or suspected hypersensitivity to ASP6294 or any components of the formulation used.
* Subject has been pregnant within 6 months prior to screening assessment or breast feeding within 3 months prior to screening.
* Subject has a known history of an allergic or anaphylactic reaction to biological drugs (e.g., [monoclonal] antibodies including tanezumab or fusion proteins).
* Subject has received a biological drug (e.g. [monoclonal] antibodies including tanezumab or fusion proteins) during the last 6 months prior to the screening visit.
* Subject has a known history of hepatitis B or C or human immunodeficiency virus (HIV) infection.
* Subject has a known history of or has a currently active or treated sexually transmittable disease (including genital herpes).
* Subject has a known current substance abuse issue (including alcoholism).
* Subject has peripheral neuropathy, or an abnormality has been observed during the sensory testing at Visit 1/Screening.
* Subject has a known currently clinically severe, unstable or uncontrolled renal, hepatic, respiratory, hematological, genitourinary (except BPS/IC), cardiovascular, endocrine, neurological, psychiatric, or other medical illness that may put the subject at safety risk or may mask measures of efficacy.
* Subject has had any malignancy diagnosed within 5 years prior to the screening visit, except for curative treated localized non-melanoma skin cancer (e.g. basal cell or squamous cell carcinoma).
* Subject has a known current psychiatric condition, mental incapacity, language barrier or the inability to read that would impair the subject's successful participation in the study.
* Subject has a body mass index of ≥ 40 kg/m^2 as sign of morbid obesity.
* Subject has any condition that makes the subject unsuitable for study participation.
* Subject has received investigational therapy (i.e., not yet approved experimental medicine) within 28 days or 5 half-lives, whichever is longer, prior to the screening visit.
* Subject is an employee of the Astellas Group, the Contract Research Organization (CRO) involved, or the investigator site executing the study.
* Results of the Visit 1/Screening blood sample indicate that the subject has active hepatic and/or biliary disease, defined as: liver enzymes aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times the upper limit of normal (ULN), or total bilirubin (TBL) > 1.5 times the ULN.
* Result of the Visit 1/Screening serum pregnancy test is positive.
* Results of the Visit 1/Screening blood/urine samples indicate that the subject has clinically significant abnormal biochemistry, hematology or urinalysis safety laboratory values.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Average Mean Daily Pain (MDP) Score at Week 12 | Baseline and Week 12
  Participants will record their MDP each day in the evening into an e-diary. The MDP is the average pain experienced over the past 24 hours. The average MDP is the mean of daily assessments of MDP in the week prior to the visit with at least 5 recordings in that week. MDP is measured using an 11-point Numerical Rating Scale (NRS) ranging from 0 (no bladder pain) to 10 (worst imaginable bladder pain). A negative change indicates a reduction/improvement from baseline.

SECONDARY OUTCOMES:
Change from Baseline in Average Worst Daily Pain (WDP) Score at Week 12 | Baseline and Week 12
  Participants will record their WDP each day in the evening into an e-diary. The WDP is the worst pain experienced over the past 24 hours. The average WDP is the mean of daily assessments of WDP in the week prior to the visit with at least 5 recordings in that week. WDP is measured using an 11-point NRS ranging from 0 (no bladder pain) to 10 (worst imaginable bladder pain). A negative change indicates a reduction/improvement from baseline.
Change From Baseline in Mean Voiding Frequency per 24 hours at Week 12 | Baseline and Week 12
  Mean voiding frequency is the mean of the recordings of voiding frequency in the electronic micturition diary in the week prior to the visit with at least 2 days recorded in that week. A negative change indicates a reduction/improvement from baseline.
Change From Baseline in Mean Number of Level 3 or 4 Urgency Episodes (Based on Patient Perception of Intensity of Urgency Scale [PPIUS]) per 24 hours at Week 12 | Baseline and Week 12
  The perceived level of urinary urgency is measured using PPIUS. For each micturition episode, participant will be asked to rate the degree of associated urgency severity according to PPIUS. PPIUS is a 5-point categorical scale ranging from 0 to 4, where 0 = no urgency (participant felt no need to empty the bladder, but did so for other reasons), 1 = mild urgency (participant could postpone voiding as long as necessary, without fear of wetting herself), 2 = moderate urgency (participant could postpone voiding for a short while, without fear of wetting herself), 3 = severe urgency (participant could not postpone voiding, had to rush to the toilet in order not to wet herself), and 4 = urge incontinence (participant leaked before arriving to the toilet). Mean number of Level 3 or 4 urgency episodes is the mean of recordings of Level 3 or 4 urgency episodes in 3-day electronic micturition diary in the week prior to visit.
Change From Baseline in Bladder Pain/ Interstitial Cystitis Symptom Score (BPIC-SS) Total Score at Week 12 | Baseline and Week 12
  The BPIC-SS is a psychometrically validated and reliable questionnaire with 8 questions concerning bladder pain over the previous 7 days. Question (Q) 1 to Q5 assess urinary symptoms (how often urinated because of pain, need to urinate just after previous urination, urination to avoid pain, pressure in the bladder, and pain in the bladder) and are rated 0 (never) to 4 (always). Q6 and Q7 assess the impact of bladder pain (bothered by frequent urination during daytime and nighttime) and are rated 0 (not at all) to 4 (a great deal). Q8 assesses the worst pain on a 0 (no bladder pain) to 10 (worst possible bladder pain) NRS. The BPIC-SS total score is the sum of the individual question scores and range from 0 to 38, with higher scores indicating a worse situation. A score of 19 or more represents moderate/severe disease activity. A negative change indicates a reduction/improvement from baseline.
Change From Baseline in BPIC-SS Worst Bladder Pain (Question 8) Score at Week 12 | Baseline and Week 12
  The BPIC-SS is a psychometrically validated and reliable questionnaire with 8 questions concerning bladder pain over the previous 7 days. Q8 of BPIC-SS assesses the worst pain on a 0 (no bladder pain) to 10 (worst possible bladder pain) NRS. A negative change indicates a reduction/improvement from baseline.
Percentage of Participants With Moderately Improved or Better Grade on the Global Response Assessment (GRA) at Week 12 | Week 12
  A self-reported 7 grade GRA is used to evaluate a participant's clinical condition relative to baseline. The GRA reads: As compared to when the participant started the study, how would the participant rate the participant's overall symptoms now? The 7 GRA grades are "markedly worse", "moderately worse", "slightly worse", "no change", "slightly improved", "moderately improved" or "markedly improved". Percentage of participants with a successful GRA response (defined as the response of "moderately improved" or better ["markedly improved"] will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Project Physician, Study Director — Astellas Pharma Europe B.V.
Locations (28):
- Site BE32001, Leuven, Belgium
- Site CZ42002, Pilsen, Czechia
- Germany (4):
  - Site DE49003, Duisburg
  - Site DE49007, Duisburg
  - Site DE49001, Holzminden
  - Site DE49005, Markkleeberg
- Hungary (2):
  - Site HU36002, Budapest
  - Site HU36001, Csongrád
- Latvia (4):
  - Site LV37103, Daugavpils
  - Site LV37101, Riga
  - Site LV37102, Riga
  - Site LV37105, Riga
- Site NL31007, Sneek, Netherlands
- Poland (4):
  - Site PL48009, Lodz
  - Site PL48002, Szczecin
  - Site PL48010, Warsaw
  - Site PL48007, Wroclaw
- Russia (5):
  - Site RU70001, Saint Petersburg
  - Site RU70002, Saint Petersburg
  - Site RU70003, Saint Petersburg
  - Site RU70006, Saint Petersburg
  - Site RU70008, Saint Petersburg
- Spain (4):
  - Site ES34001, Barcelona
  - Site ES34008, Madrid
  - Site ES34002, Málaga
  - Site ES34007, Valencia
- United Kingdom (2):
  - Site GB44002, Manchester
  - Site GB44006, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=366